CLINICAL TRIAL: NCT03973112
Title: A Single-arm, Open, Multicenter, Phase II Clinical Study Evaluating the Use of HLX10 (Recombinant Anti-pd-1 Humanized Monoclonal Antibody Injection) in Combination With HLX04 (Recombinant Anti-vegf Humanized Monoclonal Antibody Injection) for the Treatment of Advanced Hepatocellular Carcinoma (HCC) Patients
Brief Title: A Clinical Study Evaluating the Use of HLX10 in Combination With HLX04 for the Treatment of Advanced Hepatocellular Carcinoma (HCC) Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLX10-008-HCC201
Record Dates: First submitted 2019-06-02; First posted 2019-06-04 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HLX10 3 mg/kg + HLX04 5 mg/kg (Experimental): HLX10 3 mg/kg + HLX04 5 mg/kg, as second-line treatment or above
  Interventions: Drug: HLX10 3mg/kg; Drug: HLX04 5mg/kg
- HLX10 3 mg/kg + HLX04 10 mg/kg (Experimental): HLX10 3 mg/kg + HLX04 10 mg/kg,as second-line treatment or above
  Interventions: Drug: HLX10 3mg/kg; Drug: HLX04 10mg/kg
- HLX10 (Experimental): HLX10 3mg/kg, as second-line treatment or above
  Interventions: Drug: HLX10 3mg/kg
- HLX10+HLX04 1L treatment (Experimental): HLX10 3 mg/kg + HLX04 10 mg/kg: as first-line treatment
  Interventions: Drug: HLX10 3mg/kg; Drug: HLX04 10mg/kg

INTERVENTIONS:
Drug: HLX10 3mg/kg — anti-PD-1
Drug: HLX04 5mg/kg — anti-VEGF, a biosimilar to Avastin
  Arms: HLX10 3 mg/kg + HLX04 5 mg/kg
Drug: HLX04 10mg/kg — anti-VEGF, a biosimilar to Avastin
  Arms: HLX10 3 mg/kg + HLX04 10 mg/kg; HLX10+HLX04 1L treatment

SUMMARY:
This trial is a single-arm, open, multicenter phase II clinical study.Subjects can only enter this study after they meet the inclusion and exclusion criteria.Into subjects will accept HLX10 + HLX04 intravenous infusion, every two weeks, lose treatment until clinical benefit, toxicity, the subjects of the resistance or the doctor decided to suspend the treatment, tested subjects death revocation of informed consent, subjects, subjects of pregnancy, not to plan or program requirement from, or management reasons, treatment for up to 2 years (before).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet all of the following criteria are allowed to be enrolled into this study:

  * Volunteer to participate in clinical research;To fully understand and understand this study and to sign the Informed Consent Form (ICF);Willing to follow and able to complete all test procedures.
  * The age of signing ICF is ≥ 18 years old and ≤ 75 years old.
  * Subjects with advanced hepatocellular carcinoma (HCC) diagnosed by histopathology or cytology, or clinically diagnosed as meeting the criteria for hepatocellular carcinoma of the American association of liver diseases (AASLD).
  * arm A、B Failure or intolerable toxicity after at least one standard first-line systemic treatment for advanced hepatocellular carcinoma.Previous standard first-line systemic therapy included sorafenib, renvastinib and oxaliplatin based chemotherapy.
  * arm D never used systemic treatment
  * Barcelona Clinic Liver Cancer (BCLC) (appendix I) stage C;BCLC stage B patients who are not suitable for locoregional therapy may also be enrolled.
  * At least one measurable lesion assessed by IRRC according to RECIST v1.1 (appendix ii) has not been treated locally for this lesion (e.g., radiotherapy, radiofrequency ablation, TACE, ultrasound focusing knife, etc.).
  * The end of previous systematic treatment must be ≥ 2 weeks after the first medication in this study, and the treatment-related AE should be restored to the level of ci -CTCAE ≤ 1 (except hair loss).
  * Child-pugh liver function rating within 7 days before the first administration of the study drug (appendix iii) : grade A and good grade B (≤ 7 points).
  * The ECOG physical performance score (appendix iv) for the 7 days prior to the first administration of the study drug was 0 or 1.
  * Expected survival ≥ 12 weeks.
  * Subjects of HBsAg (-) and HBcAb (-) were admitted into the group;If HBsAg (+) or HBcAb (+), hbv-dna must be ≤ 500 IU/mL to be included in the group, and those with elevated hbv-dna must agree to receive nucleoside anti-hepatitis b virus treatment.Subjects with negative HCV antibody (-) or hcv-rna were admitted.If hcv-rna is positive, subjects must have ALT and AST ≤ 3×ULN to be enrolled.Subjects with co-infection of hepatitis b and c should be excluded.
  * Major organs function normally and meet the following criteria (no blood transfusion, albumin, recombinant human thrombogenin or colony stimulating factor (CSF) treatment was received within 14 days prior to the first administration of this study)
  * Female subjects must meet:

Menopause (defined as having not had menstruation for at least 1 year and having no other known cause other than menopause), or Surgical sterilization (removal of ovaries and/or uterus), or have fertility, but must meet: serum pregnancy test must be negative within 7 days prior to first administration, and , agreed to the annual failure rate < 1% of contraception or abstinence (avoid heterosexual intercourse) (from signed informed consent to test drugs at the end of the time at least 120 days) after the treatment (annual failure rate < 1% of contraceptive methods including bilateral tubal ligation, male sterilization techniques, the correct use can inhibit ovulation hormonal contracepties, releasing hormone of intrauterine contraceptive device and copper intrauterine contraceptive device), and do not breastfeed.

• Male subjects must be satisfied: agree with abstinence (avoid heterosexual intercourse) or contraceptive measures, the rules are as follows: spouse or partner has been pregnant for childbearing age women, male subjects must be at the end of the experiment during drug dosage and drug time at least 120 days after the treatment, keep abstinence or use condoms for birth control in order to prevent drug exposure in the embryo.The duration of the clinical study and the reliability of the subjects' preferences and daily lifestyle measures of abstinence should be considered.Regular abstinence (e.g., calender days, ovulation, basal body temperature, or post-ovulation methods) and ejaculation are not acceptable methods of contraception.

Exclusion Criteria:

* Subjects who meet any of the following criteria are not allowed to be enrolled in this study:

  * Hepatobiliary duct cell carcinoma, mixed cell carcinoma, or fibroblastic layer cell carcinoma are known.
  * Other active malignancies within 5 years prior to the first administration of the study drug.Curable localized tumors, such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder carcinoma, carcinoma in situ of the prostate, cervical carcinoma in situ, and carcinoma in situ of the breast, can be included in the group.
  * People who are ready to undergo or have received organ or bone marrow transplants.
  * After appropriate intervention, uncontrollable pleural effusion, pericardial effusion or ascites still need to be drained frequently (once a month or more frequently).
  * Symptomatic, untreated, or progressive central nervous system (CNS) or meningeal metastasis.Asymptomatic subjects treated for CNS lesions can be enrolled if all of the following criteria are met:

    1. in addition to CNS, there must be lesions that can be measured according to RECIST v1.1;
    2. the patient had no history of intracranial or spinal bleeding;
    3. metastatic lesions were limited to cerebellum or supratentorial areas (i.e., no mesencephalon, pons, medulla or spinal cord metastatic lesions);
    4. there was no evidence of progress between the completion of CNS oriented therapy and the start of research and treatment;
    5. the patients did not receive stereotactic radiotherapy within 7 days before the study treatment, did not receive whole-brain radiotherapy within 14 days before the study treatment, and did not receive neurosurgical resection within 28 days before the study treatment;
    6. patients have no need for continuous use of glucocorticoids in the treatment of CNS diseases.Stable doses of anticonvulsant therapy are permitted;
    7. asymptomatic patients with newly detected CNS metastases during screening are eligible to participate in the study after receiving radiotherapy or surgical treatment, and there is no need to repeat screening of brain scan results.
  * Cerebrovascular accident, myocardial infarction, unstable angina pectoris and poorly controlled arrhythmia occurred within half a year (including QTc interval ≥ 450 ms for men and ≥ 470 ms for women) (QTc interval was calculated by Fridericia formula).
  * According to the New York heart association (NYHA) standard (appendix 5) levels Ⅲ or Ⅳ cardiac insufficiency or heart colour to exceed examination: LVEF, left ventricular ejection fraction < 50%.
  * A history of hepatic encephalopathy.
  * According to the images, portal vein invasion, inferior vena cava or cardiac involvement of HCC main portal branch (Vp4) were present.Patients with cancer thrombus in main portal vein but smooth blood flow in contralateral branch can be enrolled.
  * Involving major airways, vessels, or large mediastinal mass located centrally (< 30 mm from the crest).
  * Human immunodeficiency virus (HIV) infection.
  * Active tuberculosis.
  * Patients with previous and current cases of interstitial pneumonia, pneumoconiosis, radioactive pneumonia, drug-related pneumonia, and severe impairment of lung function that may interfere with the detection and management of suspected drug-related lung toxicity.
  * Known activity or autoimmune disease or history.
  * The study drug was treated with live attenuated vaccine within 28 days prior to its first administration.
  * Subjects requiring systemic treatment with corticosteroids (> 10 mg/ day or equivalent dose of prednisone) or other immunosuppressants within 14 days prior to or during the study.In the absence of active autoimmune disease, the inhalation or topical use of steroids, or adrenal hormone replacement at doses less than 10 mg/ day of prednisone efficacy, is permitted.
  * Within 14 days prior to the first administration of the study drug, any active infection requiring systematic anti-infective treatment occurs.
  * Major surgery was performed within 28 days prior to the first administration of the study drug. Major surgery in this study was defined as the minimum recovery time of 3 weeks after surgery before the surgery treated in this study could be performed.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 2 years
  Objective response rate(assessed by independent radiological review

SECONDARY OUTCOMES:
ORR | up to 2 years
  Objective response rate (assessed by the investigators based on the RECISTv1.1
12-month OS rate | from the date of first dose unitl the date of 12-month
  12-month overall survival rate
OS | from the date of first dose unitl the date of death from any cause，assessed up to 2 years
  Overall survival (OS)
12-month PFS rate | the proportion of subjects who have time interval over 12 months between the first dose and disease progression or death
  12-month progression-free survival (PFS) rate
PFS | from the first dose until firstly confirmed and recorded disease progression or death (whichever occurs earlier),assessed up to 2 years
  Progression-free survival (assessed by independent radiological review
PFS | from the first dose until firstly confirmed and recorded disease progression or death (whichever occurs earlier),assessed up to 2 years
  Progression-free survival (assessed by the investigators based on RECIST v1.1)
DOR | from the date when CR or PR (whichever recorded earlier) is firstly achieved until the date when disease progression or death is firstly recorded (whichever occurs earlier),assessed up to 2 years
  Duration of response

CONTACTS AND LOCATIONS:
Locations (1):
- Ethics committee of zhongshan hospital affiliated to fudan university, Shanghai, China

REFERENCES:
- [Derived] Wang K, Shen Y, Hu C, Xu F, Wang Q, Gao Y, Zhou L. Population Pharmacokinetics and Exposure-Response Analysis of Serplulimab in Small Cell Lung Cancer Patients. Clin Transl Sci. 2025 Sep;18(9):e70322. doi: 10.1111/cts.70322. PMID 40932107
- [Derived] Ren Z, Shao G, Shen J, Zhang L, Zhu X, Fang W, Sun G, Bai Y, Wu J, Liu L, Yuan Y, Zhang J, Li Z, Zhang L, Yin T, Wu J, Hou X, Yu H, Li J, Wang Q, Zhu J, Fan J; Serplulimab-HCC Investigators. Phase 2 study of serplulimab with the bevacizumab biosimilar HLX04 in the first-line treatment of advanced hepatocellular carcinoma. Cancer Immunol Immunother. 2025 Jan 3;74(2):69. doi: 10.1007/s00262-024-03917-w. PMID 39751879